CLINICAL TRIAL: NCT06376695
Title: Radicle GI Health™ 24: A Randomized, Double-Blind, Placebo-Controlled, Direct-to-Consumer Study Assessing the Impact of Health and Wellness Products on Gastrointestinal (GI) Health and Related Health Outcomes
Brief Title: Radicle GI Health 24: A Study of Health and Wellness Products on GI Health and Related Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX-P-2407
Record Dates: First submitted 2024-03-28; First posted 2024-04-19 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-02

CONDITIONS: Abdominal Pain; GI Disorders; Digestion
MeSH Terms: conditions — Abdominal Pain; Digestive System Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on gender at birth then randomized to one of the study arms
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants' assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (18):
- Placebo Control 1.1 (Placebo Comparator): GI Health Product Form 1 - control
  Interventions: Dietary Supplement: Radicle GI Health Placebo Control Form 1
- Active Product 1.1 (Experimental): GI Health Product Form 1 - active product 1
  Interventions: Dietary Supplement: Radicle GI Health Active Study Product 1.1 Usage
- Placebo Control 2 (Placebo Comparator): GI Health Product Form 2 - control
  Interventions: Dietary Supplement: Radicle GI Health Placebo Control Form 2
- Active Product 2.1 (Experimental): GI Health Product Form 2 - active product 1
  Interventions: Dietary Supplement: Radicle GI Health Active Study Product 2.1 Usage
- Placebo Control 3 (Placebo Comparator): GI Health Product Form 3 - control
  Interventions: Dietary Supplement: Radicle GI Health Placebo Control Form 3
- Active Product 3.1 (Experimental): GI Health Product Form 3 - active product 1
  Interventions: Dietary Supplement: Radicle GI Health Active Study Product 3.1 Usage
- Placebo Control 4 (Placebo Comparator): GI Health Product Form 4 - control
  Interventions: Dietary Supplement: Radicle GI Health Placebo Control Form 4
- Active Product 4.1 (Experimental): GI Health Product Form 4 - active product 1
  Interventions: Dietary Supplement: Radicle GI Health Active Study Product 4.1 Usage
- Placebo Control 5 (Placebo Comparator): GI Health Product Form 5 - control
  Interventions: Dietary Supplement: Radicle GI Health Placebo Control Form 5
- Active Product 5.1 (Experimental): GI Health Product Form 5 - active product 1
  Interventions: Dietary Supplement: Radicle GI Health Active Study Product 5.1 Usage
- Placebo Control 7.1.0 (Placebo Comparator): GI Health Product Form 7.1- control
  Interventions: Dietary Supplement: Radicle GI Health Placebo Control Form 7
- Active Product 7.1.1 (Experimental): GI Health Product Form 7.1 - active product 1
  Interventions: Dietary Supplement: Radicle GI Health Active Study Product 7.1 Usage
- Placebo Control 7.2.0 (Placebo Comparator): GI Health Product Form 7.2 - control
  Interventions: Dietary Supplement: Radicle GI Health Placebo Control 7.2
- Active Product 7.2.1 (Experimental): GI Health Product Form 7.2 - active product 1
  Interventions: Dietary Supplement: Radicle GI Health Active Study Product 7.2.1 Usage
- Placebo Control 7.3.0 (Placebo Comparator): GI Health Product Form 7.3 - control
  Interventions: Dietary Supplement: Radicle GI Health Placebo Control 7.3.0
- Active Product 7.3.1 (Experimental): GI Health Product Form 7.3 - active product 1
  Interventions: Dietary Supplement: Radicle GI Health Active Study Product 7.3.1 Usage
- Placebo Control 7.4.0 (Placebo Comparator): GI Health Product Form 7.4 - control
  Interventions: Dietary Supplement: Radicle GI Health Placebo Control 7.4.0
- Active Product 7.4.1 (Experimental): GI Health Product Form 7.4 - active product 1
  Interventions: Dietary Supplement: Radicle GI Health Active Study Product 7.4.1 Usage

INTERVENTIONS:
Dietary Supplement: Radicle GI Health Placebo Control Form 1 — Participants will use their Placebo Control Form 1 as directed for a period of 6 weeks.
  Arms: Placebo Control 1.1
Dietary Supplement: Radicle GI Health Active Study Product 1.1 Usage — Participants will use their Radicle GI Health Active Study Product 1.1 as directed for a period of 6 weeks.
  Arms: Active Product 1.1
Dietary Supplement: Radicle GI Health Placebo Control Form 2 — Participants will use their Placebo Control Form 2 as directed for a period of 6 weeks.
  Arms: Placebo Control 2
Dietary Supplement: Radicle GI Health Active Study Product 2.1 Usage — Participants will use their Radicle GI Health Active Study Product 2.1 as directed for a period of 6 weeks.
  Arms: Active Product 2.1
Dietary Supplement: Radicle GI Health Placebo Control Form 3 — Participants will use their Placebo Control Form 3 as directed for a period of 6 weeks.
  Arms: Placebo Control 3
Dietary Supplement: Radicle GI Health Active Study Product 3.1 Usage — Participants will use their Radicle GI Health Active Study Product 3.1 as directed for a period of 6 weeks.
  Arms: Active Product 3.1
Dietary Supplement: Radicle GI Health Placebo Control Form 4 — Participants will use their Placebo Control Form 4 as directed for a period of 6 weeks.
  Arms: Placebo Control 4
Dietary Supplement: Radicle GI Health Active Study Product 4.1 Usage — Participants will use their Radicle GI Health Active Study Product 4.1 as directed for a period of 6 weeks.
  Arms: Active Product 4.1
Dietary Supplement: Radicle GI Health Placebo Control Form 5 — Participants will use their Placebo Control Form 5 as directed for a period of 6 weeks.
  Arms: Placebo Control 5
Dietary Supplement: Radicle GI Health Active Study Product 5.1 Usage — Participants will use their Radicle GI Health Active Study Product 5.1 as directed for a period of 6 weeks.
  Arms: Active Product 5.1
Dietary Supplement: Radicle GI Health Placebo Control Form 7 — Participants will use their Placebo Control Form 7 as directed for a period of 6 weeks.
  Arms: Placebo Control 7.1.0
Dietary Supplement: Radicle GI Health Active Study Product 7.1 Usage — Participants will use their Radicle GI Health Active Study Product 7.1 as directed for a period of 6 weeks.
  Arms: Active Product 7.1.1
Dietary Supplement: Radicle GI Health Placebo Control 7.2 — Participants will use their Placebo Control 7.2 as directed for a period of 6 weeks.
  Arms: Placebo Control 7.2.0
Dietary Supplement: Radicle GI Health Active Study Product 7.2.1 Usage — Participants will use their Radicle GI Health Active Study Product 7.2.1 as directed for a period of 6 weeks.
  Arms: Active Product 7.2.1
Dietary Supplement: Radicle GI Health Placebo Control 7.3.0 — Participants will use their Placebo Control 7.3 as directed for a period of 6 weeks.
  Arms: Placebo Control 7.3.0
Dietary Supplement: Radicle GI Health Active Study Product 7.3.1 Usage — Participants will use their Radicle GI Health Active Study Product 7.3.1 as directed for a period of 6 weeks.
  Arms: Active Product 7.3.1
Dietary Supplement: Radicle GI Health Placebo Control 7.4.0 — Participants will use their Placebo Control 7.4 as directed for a period of 6 weeks.
  Arms: Placebo Control 7.4.0
Dietary Supplement: Radicle GI Health Active Study Product 7.4.1 Usage — Participants will use their Radicle GI Health Active Study Product 7.4.1 as directed for a period of 6 weeks.
  Arms: Active Product 7.4.1

SUMMARY:
A randomized, double-blind, placebo-controlled study assessing the impact of health and wellness products on GI health and related health outcomes

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study conducted with adult participants, residing in the United States.

Eligible participants will (1) endorse a desire for improved bowel habits, less bloating/indigestion, and/or fewer stomach aches/pains (2) have the opportunity for meaningful improvement (at least 20%) in their primary health outcome, and (3) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants that report a known cardiac dysfunction, liver or kidney disease may be excluded. Participants that report a known contraindication or with well-established, significant safety concerns due to illness will be excluded. Heavy drinkers and those who report they are pregnant, trying to become pregnant, or breastfeeding will be excluded. Participants that report taking medications with a known contraindication or with well-established, significant safety concerns will be excluded.

Self-reported data are collected electronically from eligible participants for 7 weeks. Participant reports of health indicators will be collected at baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

* Adults, at least 21 years of age at the time of electronic consent, inclusive of all ethnicities, races, and gender identities. Assigned sex at birth will determine sex-specific recruitment and surveys (male vs female) employed, when needed
* Resides in the United States
* Endorses a desire for improved bowel habits, less bloating/indigestion, and/or fewer stomach aches/pains
* Has the opportunity for at least 20% improvement in their primary health outcome
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion Criteria:

* Report being pregnant, trying to become pregnant, or breastfeeding
* Unable to provide a valid US shipping address and mobile phone number
* Reports current enrollment in another clinical trial
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Reports a current and/or recent (up to 3 months ago) major illness and/or surgery that poses a known, significant safety risk.
* Reports a diagnosis of cardiac dysfunction, liver or kidney disease that presents a known contraindication and/or a significant safety risk with any of the study product ingredients. NYHA (New York Heart Association) Class Ill or IV congestive heart failure, atrial fibrillation, uncontrolled arrhythmias, cirrhosis, end-stage liver disease, stage 3b or 4 chronic kidney disease, or kidney failure
* Reports taking medications that have a well-established moderate or severe interaction, posing a substantial safety risk with any of the study product ingredients. Anticoagulants, antihypertensives, anxiolytics, antidepressants, chemotherapy, immunotherapy, sedative hypnotics, seizure medications, medications that warn against grapefruit consumption, corticosteroids at doses greater than 5 mg per day, diabetic medications, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, MAOls (monoamine oxidase inhibitors), or thyroid products
* Reports current use of the primary ingredient(s) and/or similar product(s) to the active study product(s) that may limit the effects of the study product
* Lack of reliable daily access to the internet

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4607 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Change in GI (Gastrointestinal) Health (1) | 6 weeks
  Mean difference in Gastrointestinal Health scores as assessed by Patient Reported Outcome Measurement System (PROMIS) Gastrointestinal Belly Pain 5A (scale 2-25; with higher scores corresponding to more severe abdominal pain)
Change in GI (Gastrointestinal) Health (2) | 6 weeks
  Mean difference in Gastrointestinal Health scores as assessed by Patient Reported Outcome Measurement System (PROMIS) Gastrointestinal Gas and Bloating 13A (scale 2-60; with higher scores corresponding to more severe gas/bloating)
Change in GI (Gastrointestinal) Health (3) | 6 weeks
  Mean difference in GI Health scores as assessed by Patient Reported Outcome Measurement System (PROMIS) Gastrointestinal Constipation 9A (scale 5-45; with higher scores corresponding to more severe constipation)
Change in GI (Gastrointestinal) Health (4) | 6 weeks
  Mean difference in GI Health scores as assessed by Patient Reported Outcome Measurement System (PROMIS) Gastrointestinal Diarrhea 6A (scale 2-30; with higher scores corresponding to more severe diarrhea)
Change in GI (Gastrointestinal) Health (5) | 6 weeks
  Mean difference in GI Health scores as assessed by Patient Reported Outcome Measurement System (PROMIS) Gastrointestinal Gastroesophageal Reflux 13A (scale 8-64; with higher scores corresponding to more severe reflux)
Change in GI (Gastrointestinal) Health (6) | 6 weeks
  Mean difference in GI Health scores as assessed by Patient Reported Outcome Measurement System (PROMIS) Gastrointestinal Nausea and Vomiting 4A (scale 3-20; with higher scores corresponding to more severe nausea and vomiting)

SECONDARY OUTCOMES:
Change in feelings of anxiety | 6 weeks
  Mean difference in anxiety score as assessed by PROMIS Anxiety 4A (scale 4-20; with higher scores corresponding to more severe anxiety)
Change in GI-related Quality of Life (QOL) | 6 weeks
  Mean difference in GI-related QOL as assessed by Digestion-associated QOL Questionnaire (DGLQ) (scale 0%-100%; with higher scores corresponding to worse GI-related QOL)
Change in mood (emotional distress-depression) | 6 weeks
  Mean difference in emotional distress score as assessed by PROMIS Emotional Distress- Depression 4A (scale 4-20; with higher scores corresponding to greater levels of emotional distress)
Minimal clinically important difference (MCID) in GI Health (1) | 6 weeks
  Likelihood of experiencing minimal clinically important difference in GI Health score as assessed by Patient Reported Outcome Measurement System (PROMIS) Gastrointestinal Belly Pain 5A (scale 2-25; with higher scores corresponding to more severe abdominal pain)
Minimal clinically important difference (MCID) in GI Health (2) | 6 weeks
  Likelihood of experiencing minimal clinically important difference in GI Health score as assessed by Patient Reported Outcome Measurement System (PROMIS) Gastrointestinal Gas and Bloating 13A (scale 2-60; with higher scores corresponding to more severe gas/bloating)
Minimal clinically important difference (MCID) in GI Health (3) | 6 weeks
  Likelihood of experiencing minimal clinically important difference in GI Health score as assessed by Patient Reported Outcome Measurement System (PROMIS) Gastrointestinal Constipation 9A (scale 5-45; with higher scores corresponding to more severe constipation)
Minimal clinically important difference (MCID) in GI Health (4) | 6 weeks
  Likelihood of experiencing minimal clinically important difference in GI Health score as assessed by Patient Reported Outcome Measurement System (PROMIS) Gastrointestinal Diarrhea 6A (scale 2-30; with higher scores corresponding to more severe diarrhea)
Minimal clinically important difference (MCID) in GI Health (5) | 6 weeks
  Likelihood of experiencing minimal clinically important difference in GI Health score as assessed by Patient Reported Outcome Measurement System (PROMIS) Gastrointestinal Gastroesophageal Reflux 13A (scale 8-64; with higher scores corresponding to more severe reflux)
Minimal clinically important difference (MCID) in GI Health (6) | 6 weeks
  Likelihood of experiencing minimal clinically important difference in GI Health score as assessed by Patient Reported Outcome Measurement System (PROMIS) Gastrointestinal Nausea and Vomiting 4A (scale 3-20; with higher scores corresponding to more severe nausea and vomiting)
Minimal clinically important difference (MCID) in feelings of anxiety | 6 weeks
  Likelihood of experiencing minimal clinically important difference in feelings of anxiety score as assessed by PROMIS Anxiety 4A (scale 4-20; with higher scores corresponding to more severe anxiety)
Minimal clinically important difference (MCID) in GI-related QOL | 6 weeks
  Likelihood of experiencing minimal clinically important difference in GI-related QOL score as assessed by Digestion-associated QOL Questionnaire (DGLQ) (scale 0%-100%; with higher scores corresponding to worse GI-related QOL)
Minimal clinically important difference (MCID) in mood (emotional distress-depression) | 6 weeks
  Likelihood of experiencing minimal clinically important difference in mood score as assessed by PROMIS Emotional Distress- Depression 4A (scale 4-20; with higher scores corresponding to greater levels of emotional distress)

OTHER OUTCOMES:
Change in concentration of at-home (direct-to-consumer) specimen assays either saliva, blood or stool | 6 weeks
  Mean difference in specimen assays as surrogates and/or markers for health outcomes. (Optional; among consented participants only) Potentially include saliva (IgG, cytokines, DHEA-S, Estradiol, Progesterone, Testosterone, Cortisol, Melatonin, CRP) blood (1 drop) (Cortisol, Homocysteine, Ferritin, TSH, HbA1c, Insulin, Vitamin D, DHEA-S, Testosterone, Estradiol, FSH, Total Cholesterol, HDL, LDL, Triglycerides, ApoA1, ApoB). Stool (microbial diversity). Test are optional. Unit of measure will vary based on test selected

CONTACTS AND LOCATIONS:
Overall Officials: Emily K. Pauli, PharmD, Principal Investigator — Radicle Science Inc.
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Radicle Science, Inc — http://radiclescience.com